CLINICAL TRIAL: NCT00267436
Title: Adopting and Demonstrating the Adaptation of Prevention Techniques: Community PROMISE Positives Leading and Utilizing Strategies (ADAPT CP PLUS)
Brief Title: Adopting and Demonstrating the Adaptation of Prevention Techniques: Community PROMISE PLUS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Minneapolis Urban League; (Unknown); University of Minnesota (Other); AIDS Action Committee of Massachusetts (Other); The Fenway Institute (Other)
Responsible Party: Jennifer Galbraith/ Behavioral Scientist, Centers for Disease Control and Prevention
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCHSTP-U65/CCU523908; U65/CCU523908-01
Record Dates: First submitted 2005-12-20; First posted 2005-12-21 (Estimated); Last update posted 2012-04-13 (Estimated); Status verified 2012-04

CONDITIONS: HIV Prevention; STD Prevention
Keywords: adaptation; HIV prevention; HIV positive; evidence based interventions; HIV Seronegativity
MeSH Terms: conditions — HIV Seropositivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Community PROMISE — The Community PROMISE begins with a community assessment to identify HIV risk factors. Once risk factors have been identified, individuals from the targeted at-risk community are recruited and trained to be peer advocates. Trained peer advocates interview members of the community about their behavior. Role model stories are written based on the interviews. Role model stories are personal accounts from individuals in the target population which explain how and why they took steps to practice HIV risk-reduction behaviors and the positive effects the choice has had on their lives. Each week, peer advocates distribute role model stories and supplies, such as condoms, to 10 to 20 members of their social networks.
  Other Names: AIDS Community Demonstration Project

SUMMARY:
This project will pilot test a step-by-step guide developed by CDC for organizations to engage in evidence-based adaptation of interventions previously shown to be effective in research settings for use in real world applications. The second purpose of the program is to evaluate the adapted intervention to determine if it is effective in changing behavior of HIV+ African American men who have sex with other men.

DETAILED DESCRIPTION:
During the ADAPT project both sites will adapt the original Community Promise intervention to specifically address the HIV prevention needs of sero-positive, African American men who have sex with men (HIV+ AAMSM) in either Boston, MA or Minneapolis/St. Paul (MSP), MN. The adapted intervention will be referred to as Community PROMISE, Positives Leading and Utilizing Strategies (CP PLUS).

In the first two months of the ADAPT project, the Boston and MSP sites will conduct formative evaluation activities (i.e., a comprehensive literature review, focus groups, and individual interviews) to assess the needs of the target population and organizational capacities to serve them. Results will be used to inform the adaptation of the original intervention to ensure that CP PLUS meet the expressed needs of the target population.

Process data will also be collected from various sources throughout the life of the project. Process data will be collected through staff meetings, interviews with staff, focus groups with peer advocates, and an expert panel consultation. Process data will be extremely useful for ensuring program objectives are met, improving CP PLUS, and providing information for providers in other locales who may be interested in adapting this intervention to serve this target population.

The Boston and MSP sites will also conduct outcome monitoring through collection of data concerning risk behaviors pre- and post-intervention implementation (follow-up at 6-8 months post and 11-13 months post [Boston only]) to determine if the adapted intervention has met its outcome objectives. Outcome monitoring will also be conducted for the "parent" intervention at both sites for HIV- or unknown status men who have sex with men.

In addition to the project activities, the organization will be examining the utility of the CDC draft guidance. The Boston and MSP sites are two of five case studies throughout the United States that will detail the challenges, successes and lessons learned from adapting an intervention packaged by CDC's Replicating Effective Programs (REP) and disseminated by Diffusing Effective Behavioral Interventions (DEBI) to a specific population. These findings will help other community-based organizations and Health Departments effectively adapt and tailor group, individual and community-level interventions.

ELIGIBILITY:
Inclusion Criteria:

HIV+ cohort

* Self-reports as HIV+ (for CP PLUS cohort)
* Self-report that they had sex with men in the past 3 years (MSP) or 1 year (Boston)
* Self-reports as a resident of the identified geographic areas.
* Identifies as African American
* 18 years of age, or older.

HIV- cohort

* HIV- or unknown status only, has engaged in risky sexual contact (defined as those who self-report engaging in unprotected anal or vaginal intercourse within the past year)
* Self-report that they had sex with men in the past 3 years (MSP) or 1 year (Boston)
* Identifies as African American (MSP); No racial/ethnic criteria however AA will be over-sampled and will be at least 20% of sample
* 18 years of age, or older.
* Self-reports as a resident of the identified geographic areas.
* Engage in risky sex (defined as individuals who self-report engaging in unprotected anal or vaginal intercourse within the past year.

Exclusion Criteria:

* Inability to complete informed consent process due to (a) substantial cognitive impairment. (b) non-English speaking; (c) under the influence of drugs or alcohol
* Under 18 years of age
* Plans to relocate within 12 months after baseline interview
* Anyone who does not meet inclusion criteria

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 574 (Actual)
Dates: Start 2006-07; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Sexual activities with main and casual partners in past 30 days to 6 months (i.e., unprotected insertive and receptive anal/vaginal sex and protected insertive and receptive anal/vaginal sex) | 7/2006-2/2007

SECONDARY OUTCOMES:
Behavioral intentions and attitudes for condom use; disclosure of HIV status; self reported STD diagnosis; medication adherence; links to care. | 7/2006-2/2007

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer S Galbraith, Study Director — Centers for Disease Control and Prevention
Locations (2):
- United States (2):
  - AIDS Action Committee, Boston, Massachusetts
  - Minneapolis Urban League, Minneapolis, Minnesota